CLINICAL TRIAL: NCT02415673
Title: Alignment Efficiency of Two Thermal Activated Orthodontic Archwire Sequences Based on Transition Temperature Range: A Randomized Clinical Trial
Brief Title: Alignment Efficiency of Two Thermal Activated Orthodontic Archwire Sequences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMA887599
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Crowding
Keywords: Orthodontics; Nitinol
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NiTi Af 37ºC (Experimental): Patients were treatment with fixed orthodontics appliance and arch wire. Two nickel-titanium alignment and leveling sequences were employed - NiTi archwire: 0.012 in and 0.019 X 0.025 in; and thermal activated NiTi archwires: 0.018 in and 0.016 X 0.022 in with different austenite finish temperatures (37ºC).
  Interventions: Device: Fixed orthodontics appliance and arch wire
- NiTi Af 35ºC (Experimental): Patients were treatment fixed orthodontics appliance and arch wire. Two nickel-titanium alignment and leveling sequences were employed - NiTi archwire: 0.012 in and 0.019 X 0.025 in; and thermal activated NiTi archwires: 0.018 in and 0.016 X 0.022 in with different austenite finish temperatures (35ºC)
  Interventions: Device: Fixed orthodontics appliance and arch wire

INTERVENTIONS:
Device: Fixed orthodontics appliance and arch wire — Two nickel-titanium alignment and leveling sequences were employed
  Other Names: the alignment of mandibular anterior crowding

SUMMARY:
The aim of the present study was to compare the effectiveness of two alignment sequences with thermal activated archwires with different Af temperatures applied for the correction of mandibular anterior crowding

DETAILED DESCRIPTION:
A parallel randomized clinical trial was conducted involving 42 patients ages 15 to 25 years (mean: 19.5 years) who required orthodontic treatment including the correction of mandibular anterior crowding. Eligibility criteria were no active caries, exemplary hygiene, non- extraction in the lower arch and no significant tooth size or shape abnormalities. Outcome: The primary outcome was the degree of crowding measured on plaster casts using Little's Irregularity Index. The secondary outcome was crowding survival time until the occurrence of correction in a six-month period. Randomization: The patients were randomly allocated to the different groups using sealed opaque envelopes. Blinding: The patients were blinded to the group to which they were allocated. Intervention: Patients were treatment with a pre-adjusted appliance (0.022 in- Roth prescription). Two nickel-titanium alignment and leveling sequences were employed - NiTi archwire: 0.012 in and 0.019 X 0.025 in; and thermal activated NiTi archwires: 0.018 in and 0.016 X 0.022 in with different austenite finish temperatures (37ºC and 35ºC), which formed the different study groups.

ELIGIBILITY:
Inclusion Criteria:

* Moderate mandibular anterior crowding (crowding: 4 to 6 mm) according to Little's Irregularity Index
* Presence of all teeth in lower arch through to the second molars, no indication for extractions in the lower arch
* No need for therapeutic interventions (use of inter-maxillary elastic bands, inter-dental wear, open NiTi spine, active lip bumper)
* Absence of systemic conditions that could affect tooth movements
* Absence of significant tooth size or shape abnormalities
* No history of trauma and no history of root resorption or alveolar bone loss.

Exclusion Criteria:

* Severe mandibular anterior crowding (crowding: up to 7 mm) according to Little's Irregularity Index
* Absence of any teeth in lower arch through to the second molars
* Indication for extractions in the lower arch
* Need for therapeutic interventions (use of inter-maxillary elastic bands, inter-dental wear, open NiTi spine, active lip bumper)
* Presence of systemic conditions that could affect tooth movements
* Presence of significant tooth size or shape abnormalities
* History of trauma and history of root resorption or alveolar bone loss.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2010-08; Primary Completion 2011-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Degree of crowding measured on plaster casts using Little's Irregularity Index | 6 months

SECONDARY OUTCOMES:
crowding survival time | six months